CLINICAL TRIAL: NCT02479737
Title: The Active Clearance Technology (ACT) II German Multicenter Trial
Brief Title: Active Clearance Technology (ACT) II German Multicenter Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Dr. Theodor Fischlein (Other)
Collaborators: ClearFlow, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Theodor Fischlein, Head, Department of Cardiac Surgery, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Other Study IDs: Germany-ACT II
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Heart Surgery
Keywords: Chest tube; chest drainage; retained blood complications; chest tube clogging; hemothorax; tamponade; heart surgery; pleural effusion; intensive care
MeSH Terms: conditions — Hemothorax; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Blood drainage post cardiac surgery using PleuraFlow System

SUMMARY:
Postoperative bleeding is a common consequence after heart surgery which can significantly impact outcomes and costs [Wynne R, Christensen MC, Dixon B]. When bleeding occurs, reliable postoperative blood evacuation of the pleural, mediastinal and pericardial spaces with chest tubes is imperative to facilitate pulmonary re-expansion and mediastinal decompression as the patient recovers. When postoperative blood evacuation is inadequate, retained blood complications can result (herein described as the Retained Blood Complications (RBC). RBC is the presence of post-operative pericardial and/or pleural fluid or blood that is diagnosed and may necessitate drainage in the acute or sub-acute setting. The need for treatment and interventions for these conditions represents an impediment to patient recovery and involves both resource and economic consumption for a heart program and the healthcare system at large.

Clinically, Retained Blood Complications (RBC) can be recognized acutely or subacutely. When it presents acutely, it is usually fresh thrombus around the heart or lungs presenting as tamponade or hemothorax. When it presents subacutely, it results in bloody pleural or pericardial effusions. These effusions are often driven by the breakdown of remaining thrombus. Once RBC occurs, subsequent procedures may be needed to remedy it.

A recent review of the literature indicated that additional procedures for RBC are demonstrated in approximately 15% to 20% of patients after heart surgery. In a prospectively collected United States Nationwide Inpatient Sample (NIS) data from 2010, RBC could be demonstrated in 17% of patients. In this analysis, mortality was doubled from 4% to 8%, length of stay was increased by 5 days, and average costs were 55% higher. Patients with RBC, therefore, represent an increased at risk population for complications and costs.

Postoperative obstruction of conventional chest tubes with blood and other fibrinous material in the setting of postoperative bleeding contributes to RBC. (Shalli) In a recent study of postoperative cardiac surgery patients at the Cleveland Clinic, 36% of patients were found to have evidence of chest tube obstruction . Active Clearance with PleuraFlow has been shown to prevent chest tube clogging, and reduce RBC.

DETAILED DESCRIPTION:
Complications from RBS are defined as those requiring re-operation or surgical interventions to evacuate blood, blood clot, bloody fluid, and air accumulation within the operative site after closure of the surgical wound. This is a prospective multicenter observational post-market study with a retrospective component. The study is open to up to five (5) German sites enrolling a consecutive cohort of cardiac surgery patients.

There are two conditions for participation in this registry. First, sites are required to enter into the study database anonymized matched historical data elements from a cohort of cardiac surgery patients done over the preceding 12 to 24-month period (Phase 0). These retrospective data elements will be used as baseline information for the purpose of comparative analyses with the prospective data sets. Second, sites that have not been using the PleuraFlow System before enrolling patients to this study are required to participate in a roll-in phase (Phase 1). The purposes of the roll-in phase are to allow the users at participating sites to familiarize themselves with the product use and with ACT, to implement Clinical Use Protocols provided by ClearFlow, Inc. to all commercial users as part of product training, and to demonstrate consistency and compliance with the clinical use protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects 18 years or older who received a PleuraFlow System following heart surgery

Exclusion Criteria:

1. Any condition deemed inappropriate for inclusion by the investigators
2. Infants, children and adolescents under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects older than 18 years who received a PleuraFlow System following heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 1113 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in the rate of interventions to treat Retained Blood Syndrome (RBS) | participants will be followed for the duration of hospital stay, an expected average of 12 days
  RBS is a composite endpoint defined as an intervention to treat one or more of the following conditions:
  -Re-exploration for bleeding, tamponade or washout of retained bloo

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Fischlein, Prof., Principal Investigator — Paracelsus Medical University, Klinikum, Nuremberg, Germany
Locations (2):
- Germany (2):
  - Herz- und Gefäßklinik GmbH, Bad Neustadt an der Saale, Bavaria
  - Paracelsus Medical University, Klinikum, Nuremberg, Germany, Nuremberg, Bavaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wynne R, Botti M, Copley D, Bailey M. The normative distribution of chest tube drainage volume after coronary artery bypass grafting. Heart Lung. 2007 Jan-Feb;36(1):35-42. doi: 10.1016/j.hrtlng.2006.05.006. PMID 17234475
- [Background] Christensen MC, Dziewior F, Kempel A, von Heymann C. Increased chest tube drainage is independently associated with adverse outcome after cardiac surgery. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):46-51. doi: 10.1053/j.jvca.2011.09.021. Epub 2011 Nov 18. PMID 22100857
- [Background] Dixon B, Santamaria JD, Reid D, Collins M, Rechnitzer T, Newcomb AE, Nixon I, Yii M, Rosalion A, Campbell DJ. The association of blood transfusion with mortality after cardiac surgery: cause or confounding? (CME). Transfusion. 2013 Jan;53(1):19-27. doi: 10.1111/j.1537-2995.2012.03697.x. Epub 2012 May 11. PMID 22574710
- [Background] Light RW. Pleural effusions following cardiac injury and coronary artery bypass graft surgery. Semin Respir Crit Care Med. 2001 Dec;22(6):657-64. doi: 10.1055/s-2001-18802. PMID 16088710
- [Background] Light RW. Pleural effusions after coronary artery bypass graft surgery. Curr Opin Pulm Med. 2002 Jul;8(4):308-11. doi: 10.1097/00063198-200207000-00011. PMID 12055394
- [Background] Light RW, Rogers JT, Cheng D, Rodriguez RM. Large pleural effusions occurring after coronary artery bypass grafting. Cardiovascular Surgery Associates, PC. Ann Intern Med. 1999 Jun 1;130(11):891-6. doi: 10.7326/0003-4819-130-11-199906010-00004. PMID 10375337
- [Background] Light RW, Rogers JT, Moyers JP, Lee YC, Rodriguez RM, Alford WC Jr, Ball SK, Burrus GR, Coltharp WH, Glassford DM Jr, Hoff SJ, Lea JW 4th, Nesbitt JC, Petracek MR, Starkey TD, Stoney WS, Tedder M. Prevalence and clinical course of pleural effusions at 30 days after coronary artery and cardiac surgery. Am J Respir Crit Care Med. 2002 Dec 15;166(12 Pt 1):1567-71. doi: 10.1164/rccm.200203-184OC. Epub 2002 Oct 11. PMID 12406850
- [Background] Ikaheimo MJ, Huikuri HV, Airaksinen KE, Korhonen UR, Linnaluoto MK, Tarkka MR, Takkunen JT. Pericardial effusion after cardiac surgery: incidence, relation to the type of surgery, antithrombotic therapy, and early coronary bypass graft patency. Am Heart J. 1988 Jul;116(1 Pt 1):97-102. doi: 10.1016/0002-8703(88)90255-4. PMID 3260740
- [Background] Clark G, Licker M, Bertin D, Spiliopoulos A. Small size new silastic drains: life-threatening hypovolemic shock after thoracic surgery associated with a non-functioning chest tube. Eur J Cardiothorac Surg. 2007 Mar;31(3):566-8. doi: 10.1016/j.ejcts.2006.12.010. Epub 2007 Jan 9. PMID 17215136
- [Background] Karimov JH, Gillinov AM, Schenck L, Cook M, Kosty Sweeney D, Boyle EM, Fukamachi K. Incidence of chest tube clogging after cardiac surgery: a single-centre prospective observational study. Eur J Cardiothorac Surg. 2013 Dec;44(6):1029-36. doi: 10.1093/ejcts/ezt140. Epub 2013 Mar 21. PMID 23520232
- [Background] Shalli S, Boyle EM, Saeed D, Fukamachi K, Cohn WE, Gillinov AM. The active tube clearance system: a novel bedside chest-tube clearance device. Innovations (Phila). 2010 Jan;5(1):42-7. doi: 10.1097/IMI.0b013e3181cf7ce3. PMID 22437275
- [Background] Shiose A, Takaseya T, Fumoto H, Arakawa Y, Horai T, Boyle EM, Gillinov AM, Fukamachi K. Improved drainage with active chest tube clearance. Interact Cardiovasc Thorac Surg. 2010 May;10(5):685-8. doi: 10.1510/icvts.2009.229393. Epub 2010 Feb 23. PMID 20179137
- [Background] Arakawa Y, Shiose A, Takaseya T, Fumoto H, Kim HI, Boyle EM, Gillinov AM, Fukamachi K. Superior chest drainage with an active tube clearance system: evaluation of a downsized chest tube. Ann Thorac Surg. 2011 Feb;91(2):580-3. doi: 10.1016/j.athoracsur.2010.10.018. PMID 21256318
- [Background] Perrault LP, Pellerin M, Carrier M, Cartier R, Bouchard D, Demers P, Boyle EM. The PleuraFlow Active Chest Tube Clearance System: initial clinical experience in adult cardiac surgery. Innovations (Phila). 2012 Sep-Oct;7(5):354-8. doi: 10.1097/IMI.0b013e31827e2b4d. PMID 23274869